CLINICAL TRIAL: NCT07398976
Title: Sex Differences in E-Cigarette Perception: Study 2
Brief Title: Sex Differences in E-Cigarette Perception
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000041248; 5K01DA056494 (NIH)
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Nicotine Dependence; E-cigarette Use
Keywords: Sex Differences; Females; E-cigarettes; Menthol; Nicotine; Vaping
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Intervention Model Description: Study is a within subject design. All participants are exposed to the same three e-liquids in randomized order under double-blinded conditions in the Lab 1 sampling session. In Lab 2, two of the three e-liquids (the same two across participants) are tested in a concurrent choice session.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will test three e-cigarettes in containing varying levels of nicotine and menthol in a sampling session in Lab 1 in a double blinded randomized order. Investigator and research assistant (i.e., care provider) will know the nicotine concentrations and menthol level of the three e-cigarettes, but will be blinded to the order of presentation/participant.
  For Lab 2, two of the three e-cigarettes are compared in a choice task. The participant will not know the nicotine or menthol of the e-cigarettes (but as they will be labeled the same as Lab 1, so will have prior experience with them). The investigator and research assistant will know the e-cigarettes as a function of the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sampling Session - Lab 1 (Experimental): Participants will sample and rate three menthol flavored e-cigarettes with varying levels of nicotine.
  Interventions: Other: Nicotine Level 1 (0mg/ml); Other: Nicotine Level 2 (36mg/ml); Other: Nicotine Level 3 (59mg/ml)
- Concurrent Choice Session- Lab 2 (Experimental): Participants will make choices between two menthol e-cigarettes with different levels of nicotine.
  Interventions: Other: Nicotine Level 1 (0mg/ml); Other: Nicotine Level 2 (36mg/ml)

INTERVENTIONS:
Other: Nicotine Level 1 (0mg/ml) — Menthol with be paired with 0mg/ml nicotine in an e-cigarette
Other: Nicotine Level 2 (36mg/ml) — Menthol with be paired with 36mg/ml nicotine in an e-cigarette
Other: Nicotine Level 3 (59mg/ml) — Menthol with be paired with 59mg/ml nicotine in an e-cigarette
  Arms: Sampling Session - Lab 1

SUMMARY:
This study examines differences between males and females in the appeal and addiction potential of menthol flavored e-cigarettes with and without nicotine.

DETAILED DESCRIPTION:
The goal of this protocol is to investigate how sex differences in response to menthol and nicotine influence product preference and choice. In this proposal, participants will be exposed to menthol non-nicotine and nicotine containing e-cigarettes and product preference and choice will be examined in a paradigm where a menthol nicotine-containing e-cigarette is progressively more difficult to earn, and a menthol non-nicotine e-cigarette is available at a low, fixed cost. Additionally, it will be investigated how menthol e-cigarettes with and without nicotine impact reward, appeal, and sensory effects in an initial sampling session (secondary and exploratory outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Able to read/write in English
* Current cigarette smoking
* Prior e-cigarette exposure
* Biochemically verified cigarette use
* Not trying to quit tobacco use

Exclusion Criteria:

* Significant medical concerns that would increase study risk
* Use of psychoactive drugs unless prescribed and stable
* Allergy to menthol or other e-liquid ingredients
* Dislike of menthol
* Pregnant, trying to get pregnant, breastfeeding

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Choices | For the 3 hour period of the Lab 2 preference task
  Differences in proportion of choices for the two menthol e-cigarette for males and females in the Lab 2 preference task
Breakpoint | During the 3 hour period of the Lab 2 preference task
  Difference in highest point of the progressive ratio schedule obtained between males and females

SECONDARY OUTCOMES:
Reward | Immediately (~2 minutes) after e-cigarette exposures in Lab 1
  Difference in scores (range: 0-100) of the Liking/Wanting Subscale of the Drug Effects Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Danielle R Davis, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigator may share information about the IPD and study results with other researchers in the future, but the information will be de-identified.
Supporting Information: ICF
Access Criteria: The de-identified data may be made available for research purposes after study publication by contacting the PI.